CLINICAL TRIAL: NCT03993574
Title: Feasibility of a Stroke Specific Self-management Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH); The Claude D. Pepper Older Americans Independence Centers (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 19-0006
Record Dates: First submitted 2019-06-18; First posted 2019-06-20 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-09

CONDITIONS: Stroke; Chronic Conditions
MeSH Terms: conditions — Stroke; Chronic Disease | interventions — Self-Management; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (Other): The standard care group will receive baseline testing #1, standard care, baseline testing #2 and follow up testing approximately 8 weeks later.
  Interventions: Other: Standard care
- Experimental (Experimental): Experimental group will baseline testing #1, standard care, baseline testing #2 however then participate in a 6-week self-management intervention (either generic or vision specific self-management based) and then get 8 week follow up testing.
  Interventions: Other: Self- management program

INTERVENTIONS:
Other: Self- management program — The program sessions are either adapted from the Stanford Patient Education Research Center's program called the Chronic Disease Self-Management Program (CDSMP) or from a vision self-management program.
  Despite which self-management program, the format for each session will include, review of educational materials (using the CDSMP book/article), discussion via a case vignette (which is always stroke related), and participation in an activity based on that session's topic. These group sessions will be 1.5 hours each week for 6 weeks
  Arms: Experimental
Other: Standard care — All stroke patients being discharged from the acute hospital receive the following care:
  1. 1 follow-up call within 2 weeks by a nurse coordinator. The call involves checking if medications were able to be filled and how the person is feeling.
  2. A stroke clinic appointment that is set to occur 90-days post discharge.
  3. A list of their personal medications and generic educational materials. The educational materials are standard forms located in the Epic system. It is the nurses' responsibility to choose what forms to provide, however it is mandatory that stroke risk factor information is included.
  4. Information on local support groups.
  5. Referrals to start physical, occupational or speech therapy, if recommended by their physician.
  Arms: Standard Care

SUMMARY:
Stroke is a leading cause of disability, institutionalization, readmission and death. This research is being completed to accelerate the adoption of evidence-based therapy practices that improve overall stroke care and outcomes. We will implement a feasibility randomized controlled trial (RCT) studying the implementation of a stroke specific chronic disease self-management program. Specifically, if the person is identified to have a chronic vision impairment identified on the vision screen, a specific low vision self-management program will be used. Otherwise the program that will be used is the generic chronic disease self-management program.

DETAILED DESCRIPTION:
Approximately 75% of people are living with a prevalent chronic disease like diabetes or hypertension. Despite this high percentage, there is a projected increase of 37% by 2030. There are approximately 795,000 people sustaining a stroke each year, in the United States. Surviving a stroke can cost an estimated $34 billion dollars a year in medical costs and loss of productivity. While there is a sharp decline in mortality rate following stroke, the rate of long-term residual impairments, disabilities and risk for developing high rates of secondary chronic conditions remains high. People living with a new stroke can also have chronic conditions in their past medical histories. Management of prior and new conditions may not become evident until the stroke survivor has returned to the community and are no longer receiving medical services. Additionally, management of chronic conditions, especially for people who now are recovering from a stroke, may require different management plans altogether. The Center for Disease Control and Prevention called for a public health action to address chronic illness. One type of community rehabilitation intervention method is self-management.

Self-management was first developed for well-elderly with chronic diseases. These programs support individuals managing their independently managing symptoms as well as help with the emotional and physical stress associated with chronic disease. Multiple research reports conclude that self-management interventions improve health outcomes, help with management of self-identity and reduce health care costs.

There are existing stroke specific self-management programs, however minimal reported research regarding the best way to implement and measure a stroke specific chronic disease self-management program to optimize health outcomes and improve quality of life. Recently, a qualitative study concluded that any stroke specific self-management program should include 3 conceptual layers to address individual, external and environmental factors essential to enable successful implementation. The first conceptual layer is individual capacity or readiness to respond to the demands to self-management. The second is having external support for self-management. And the third is being in an environment that supports and facilitates success. Another study reported strong feasibility evidence for stroke specific self-management programs versus a standard program for community dwelling stroke survivors. A small study reported a program administered to stroke patients that led to changes in self-efficacy.

Consistent with a feasibility study for implementing evidence based intervention, this project intends to address a need to bridge the translation gap between research evidence and clinical practice. This project intends to provide information to add to existing literature regarding implementation. Thus we plan to use the Determinant Framework, which will help specify determinants which act as barriers and enablers that influence implementation outcomes. Additionally, implementation theories will help us assess the implementation context, as we plan to use a checklist to evaluate factors influencing implementation across different domains (e.g. fidelity). This study also intends to provide preliminary data regarding efficacy in order to determine if a stroke specific program was superior to standard care.

ELIGIBILITY:
Inclusion Criteria:

* Acute hospitalization due to diagnosis of stroke
* at least one chronic medical condition
* must be able to consent independently
* be alert and oriented x 3
* be ≥ 18 years old

Exclusion Criteria:

* unable to independently consent
* they do not speak English
* discharged from acute care to nursing home

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility: Patients Screened | Collected at baseline 1 (24 hours prior to the patients' discharge from acute care)
  number of patients screened
Feasibility: Eligible Patients | Collected at baseline 1 (24 hours prior to the patients' discharge from acute care)
  number of patients eligible
Feasibility: Patients Approached | Collected at baseline 1 (24 hours prior to the patients' discharge from acute care)
  number of patients approached
Feasibility: Patients Enrolled | Collected at baseline 1 (24 hours prior to the patients' discharge from acute care)
  number of patients enrolled
Feasibility: Patient Refusals | Collected at follow-up (2 weeks from last day of intervention)
  number of patient refusals
Feasibility: Patient Withdrawals | Collected at follow-up (2 weeks from last day of intervention)
  number of patient withdrawals

SECONDARY OUTCOMES:
Change in self-reported self-management, as measured by the Southampton Stroke Self-Management Questionnaire | change in self- management from base line 1 (24 hours prior to discharge from acute care) to base line 2 (3 months)
  patient-reported outcome measure (PROM) of self-management competency following stroke, likert scale 1-6, higher scores on the scale equal less self-management skills
Change in self-reported self-management, as measured by the Southampton Stroke Self-Management Questionnaire | change in self-management from base line 2 (3 months) to follow-up (2 weeks from last day of intervention)
  patient-reported outcome measure (PROM) of self-management competency following stroke, likert scale 1-6, higher scores on the scale equal less self-management skills
Change in self-reported self-efficacy, as measured by the Patient Reported Outcome Measure Information System (PROMIS) self-efficacy scale | change in self-efficacy from base line 1 (24 hours prior to discharge from acute care), base line 2 (3 months)
  Self-Efficacy for Managing: Daily Activities, Symptoms, Medications and Treatments, Emotions, and Social Interactions. Likert scale 1-5, higher scores on the scale equal better confidence
Change in self-reported self-efficacy, as measured by the Patient Reported Outcome Measure Information System (PROMIS) self-efficacy scale | change in self-efficacy from base line 2 (3 months) to follow-up (2 weeks from last day of intervention)
  Self-Efficacy for Managing: Daily Activities, Symptoms, Medications and Treatments, Emotions, and Social Interactions. Likert scale 1-5, higher scores on the scale equal better confidence
Change in self-reported sleep, as measured by the PROMIS sleep disturbance and sleep-related impairments | change in sleep from base line 1 (24 hours prior to discharge from acute care), base line 2 (3 months)
  qualitative aspects of sleep and wake function via Likert scale of 1-5, higher scores on the scale equal better sleep
Change in self-reported sleep, as measured by the PROMIS sleep disturbance and sleep-related impairments | change in sleep from base line 2 (3 months) to follow-up (2 weeks from last day of intervention)
  qualitative aspects of sleep and wake function via Likert scale of 1-5, higher scores on the scale equal better sleep
Change in self-reported vision, as measured by the national eye institute vision function questionnaire -25 | change in vision quality of life from base line 1 (24 hours prior to discharge from acute care) to base line 2 (3 months)
  vision quality of life, likert scale 1-5, higher scores on the scale equal better visual function
Change in self-reported vision, as measured by the national eye institute vision function questionnaire -25 | change in vision quality of life from base line 2 (3 months) to follow-up (2 weeks from last day of intervention)
  vision quality of life, likert scale 1-5, higher scores on the scale equal better visual function

OTHER OUTCOMES:
Change in self-reported health distress, as measured by the Health Distress Questionnaire | change in health distress from base line 1 (24 hours prior to discharge from acute care) to base line 2 (3 months)
  health distress, likert scale 0-5, higher scores on the scale equal more distress.
Change in self-reported health distress, as measured by the Health Distress Questionnaire | change in health distress from base line 2 (3 months) to follow-up (2 weeks from last day of intervention)
  health distress, likert scale 0-5, higher scores on the scale equal more distress.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Reistetter, PhD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benjamin EJ, Blaha MJ, Chiuve SE, Cushman M, Das SR, Deo R, de Ferranti SD, Floyd J, Fornage M, Gillespie C, Isasi CR, Jimenez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Mackey RH, Matsushita K, Mozaffarian D, Mussolino ME, Nasir K, Neumar RW, Palaniappan L, Pandey DK, Thiagarajan RR, Reeves MJ, Ritchey M, Rodriguez CJ, Roth GA, Rosamond WD, Sasson C, Towfighi A, Tsao CW, Turner MB, Virani SS, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS, Muntner P; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2017 Update: A Report From the American Heart Association. Circulation. 2017 Mar 7;135(10):e146-e603. doi: 10.1161/CIR.0000000000000485. Epub 2017 Jan 25. No abstract available. Erratum In: Circulation. 2017 Mar 7;135(10):e646. doi: 10.1161/CIR.0000000000000491. Circulation. 2017 Sep 5;136(10):e196. doi: 10.1161/CIR.0000000000000530. PMID 28122885
- [Background] Yang Q, Tong X, Schieb L, Vaughan A, Gillespie C, Wiltz JL, King SC, Odom E, Merritt R, Hong Y, George MG. Vital Signs: Recent Trends in Stroke Death Rates - United States, 2000-2015. MMWR Morb Mortal Wkly Rep. 2017 Sep 8;66(35):933-939. doi: 10.15585/mmwr.mm6635e1. PMID 28880858
- [Background] Proctor E, Silmere H, Raghavan R, Hovmand P, Aarons G, Bunger A, Griffey R, Hensley M. Outcomes for implementation research: conceptual distinctions, measurement challenges, and research agenda. Adm Policy Ment Health. 2011 Mar;38(2):65-76. doi: 10.1007/s10488-010-0319-7. PMID 20957426
- [Background] Bowen DJ, Kreuter M, Spring B, Cofta-Woerpel L, Linnan L, Weiner D, Bakken S, Kaplan CP, Squiers L, Fabrizio C, Fernandez M. How we design feasibility studies. Am J Prev Med. 2009 May;36(5):452-7. doi: 10.1016/j.amepre.2009.02.002. PMID 19362699
- [Background] Boger EJ, Hankins M, Demain SH, Latter SM. Development and psychometric evaluation of a new patient -reported outcome measure for stroke self -management: The Southampton Stroke Self - Management Questionnaire (SSSMQ). Health Qual Life Outcomes. 2015 Oct 3;13:165. doi: 10.1186/s12955-015-0349-7. PMID 26432093
- [Background] Gruber-Baldini AL, Velozo C, Romero S, Shulman LM. Validation of the PROMIS(R) measures of self-efficacy for managing chronic conditions. Qual Life Res. 2017 Jul;26(7):1915-1924. doi: 10.1007/s11136-017-1527-3. Epub 2017 Feb 26. PMID 28239781
- [Background] Buysse DJ, Yu L, Moul DE, Germain A, Stover A, Dodds NE, Johnston KL, Shablesky-Cade MA, Pilkonis PA. Development and validation of patient-reported outcome measures for sleep disturbance and sleep-related impairments. Sleep. 2010 Jun;33(6):781-92. doi: 10.1093/sleep/33.6.781. PMID 20550019
- [Background] Rine RM, Roberts D, Corbin BA, McKean-Cowdin R, Varma R, Beaumont J, Slotkin J, Schubert MC. New portable tool to screen vestibular and visual function--National Institutes of Health Toolbox initiative. J Rehabil Res Dev. 2012;49(2):209-20. doi: 10.1682/jrrd.2010.12.0239. PMID 22773523
- [Background] Lorig K, Stewart A, Ritter P, González V, et al. Outcome Measures for Health Education and Other Health Care Interventions. Thousand Oaks, CA, US: Sage Publications, Inc; 1996.
- [Background] Harris JR, Wallace RB. The Institute of Medicine's new report on living well with chronic illness. Prev Chronic Dis. 2012;9:E148. doi: 10.5888/pcd9.120126. No abstract available. PMID 22995102
- [Background] Mozaffarian D, Benjamin EJ, Go AS, Arnett DK, Blaha MJ, Cushman M, de Ferranti S, Despres JP, Fullerton HJ, Howard VJ, Huffman MD, Judd SE, Kissela BM, Lackland DT, Lichtman JH, Lisabeth LD, Liu S, Mackey RH, Matchar DB, McGuire DK, Mohler ER 3rd, Moy CS, Muntner P, Mussolino ME, Nasir K, Neumar RW, Nichol G, Palaniappan L, Pandey DK, Reeves MJ, Rodriguez CJ, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Willey JZ, Woo D, Yeh RW, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2015 update: a report from the American Heart Association. Circulation. 2015 Jan 27;131(4):e29-322. doi: 10.1161/CIR.0000000000000152. Epub 2014 Dec 17. No abstract available. PMID 25520374
- [Background] Laver K, Halbert J, Stewart M, Crotty M. Patient readiness and ability to set recovery goals during the first 6 months after stroke. J Allied Health. 2010 Winter;39(4):e149-54. PMID 21184017
- [Background] Gallacher K, Morrison D, Jani B, Macdonald S, May CR, Montori VM, Erwin PJ, Batty GD, Eton DT, Langhorne P, Mair FS. Uncovering treatment burden as a key concept for stroke care: a systematic review of qualitative research. PLoS Med. 2013;10(6):e1001473. doi: 10.1371/journal.pmed.1001473. Epub 2013 Jun 25. PMID 23824703
- [Background] Allen K, Hazelett S, Jarjoura D, Wright KD, Clough L, Weinhardt J. Improving stroke outcomes: Implementation of a postdischarge care management model. J Clin Outcomes Manag. 2004;11(11):707-714.
- [Background] Smith ML, Ory MG, Ahn S, Kulinski KP, Jiang L, Horel S, Lorig K. National dissemination of chronic disease self-management education programs: an incremental examination of delivery characteristics. Front Public Health. 2015 Apr 27;2:227. doi: 10.3389/fpubh.2014.00227. eCollection 2014. PMID 25964923
- [Background] Lorig KR, Ritter P, Stewart AL, Sobel DS, Brown BW Jr, Bandura A, Gonzalez VM, Laurent DD, Holman HR. Chronic disease self-management program: 2-year health status and health care utilization outcomes. Med Care. 2001 Nov;39(11):1217-23. doi: 10.1097/00005650-200111000-00008. PMID 11606875
- [Background] Lorig KR, Holman H. Self-management education: history, definition, outcomes, and mechanisms. Ann Behav Med. 2003 Aug;26(1):1-7. doi: 10.1207/S15324796ABM2601_01. PMID 12867348
- [Background] Lorig KR, Sobel DS, Stewart AL, Brown BW Jr, Bandura A, Ritter P, Gonzalez VM, Laurent DD, Holman HR. Evidence suggesting that a chronic disease self-management program can improve health status while reducing hospitalization: a randomized trial. Med Care. 1999 Jan;37(1):5-14. doi: 10.1097/00005650-199901000-00003. PMID 10413387
- [Background] Jones F, Riazi A. Self-efficacy and self-management after stroke: a systematic review. Disabil Rehabil. 2011;33(10):797-810. doi: 10.3109/09638288.2010.511415. Epub 2010 Aug 27. PMID 20795919
- [Background] Kralik D, Koch T, Price K, Howard N. Chronic illness self-management: taking action to create order. J Clin Nurs. 2004 Feb;13(2):259-67. doi: 10.1046/j.1365-2702.2003.00826.x. PMID 14723679
- [Background] Ahn S, Basu R, Smith ML, Jiang L, Lorig K, Whitelaw N, Ory MG. The impact of chronic disease self-management programs: healthcare savings through a community-based intervention. BMC Public Health. 2013 Dec 6;13:1141. doi: 10.1186/1471-2458-13-1141. PMID 24314032
- [Background] Boger EJ, Demain S, Latter S. Self-management: a systematic review of outcome measures adopted in self-management interventions for stroke. Disabil Rehabil. 2013 Aug;35(17):1415-28. doi: 10.3109/09638288.2012.737080. Epub 2012 Nov 21. PMID 23167558
- [Background] Jones F, Mandy A, Partridge C. Changing self-efficacy in individuals following a first time stroke: preliminary study of a novel self-management intervention. Clin Rehabil. 2009 Jun;23(6):522-33. doi: 10.1177/0269215508101749. Epub 2009 Apr 29. PMID 19403556
- [Background] Harwood M, Weatherall M, Talemaitoga A, Barber PA, Gommans J, Taylor W, McPherson K, McNaughton H. Taking charge after stroke: promoting self-directed rehabilitation to improve quality of life--a randomized controlled trial. Clin Rehabil. 2012 Jun;26(6):493-501. doi: 10.1177/0269215511426017. Epub 2011 Nov 15. PMID 22087047
- [Background] Boger EJ, Demain SH, Latter SM. Stroke self-management: a focus group study to identify the factors influencing self-management following stroke. Int J Nurs Stud. 2015 Jan;52(1):175-87. doi: 10.1016/j.ijnurstu.2014.05.006. Epub 2014 May 24. PMID 24917370
- [Background] Battersby M, Hoffmann S, Cadilhac D, Osborne R, Lalor E, Lindley R. 'Getting your life back on track after stroke': a Phase II multi-centered, single-blind, randomized, controlled trial of the Stroke Self-Management Program vs. the Stanford Chronic Condition Self-Management Program or standard care in stroke survivors. Int J Stroke. 2009 Apr;4(2):137-44. doi: 10.1111/j.1747-4949.2009.00261.x. PMID 19383056
- [Background] Cadilhac DA, Hoffmann S, Kilkenny M, Lindley R, Lalor E, Osborne RH, Batterbsy M. A phase II multicentered, single-blind, randomized, controlled trial of the stroke self-management program. Stroke. 2011 Jun;42(6):1673-9. doi: 10.1161/STROKEAHA.110.601997. Epub 2011 Apr 14. PMID 21493910
- [Background] Nilsen P. Making sense of implementation theories, models and frameworks. Implement Sci. 2015 Apr 21;10:53. doi: 10.1186/s13012-015-0242-0. PMID 25895742
- [Background] Carroll C, Patterson M, Wood S, Booth A, Rick J, Balain S. A conceptual framework for implementation fidelity. Implement Sci. 2007 Nov 30;2:40. doi: 10.1186/1748-5908-2-40. PMID 18053122
- [Background] Living a Healthy Life with Chronic Conditions, 4th Edition. https://www.bullpub.com/living-a-healthy-life-with-chronic-conditions-4th-edition.html
- [Background] Rees G, Keeffe JE, Hassell J, Larizza M, Lamoureux E. A self-management program for low vision: program overview and pilot evaluation. Disabil Rehabil. 2010;32(10):808-15. doi: 10.3109/09638280903304193. PMID 20367406